CLINICAL TRIAL: NCT00676416
Title: Influence of Propofol on Alveolar Macrophage Immunity in Asthmatic Patients Undergoing General Anesthesia
Brief Title: Influence of Propofol on Alveolar Macrophage in Asthmatic Patients
Acronym: PAMAP
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: HRSA/Maternal and Child Health Bureau (U.S. Federal Agency)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Other Study IDs: NMCHCH-0288-323; NMU-08-1090
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Asthma
Keywords: General anesthesia; Propofol; Immunity; Alveolar Macrophages
MeSH Terms: conditions — Asthma | interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Propofol general anesthesia for asthmatic patients
  Interventions: Drug: 2,6-Diisopropylphenol
- 2: Propofol general anesthesia for non-asthmatic patients
  Interventions: Drug: 2,6-Diisopropylphenol

INTERVENTIONS:
Drug: 2,6-Diisopropylphenol — Propofol general anesthesia was performed in patients with asthma (1) and without asthma (2)
  Other Names: Diprivan

SUMMARY:
The change of airway responsiveness and alveolar macrophage (AM) immunity occurs during the pathogenesis of asthma. Macrophage-associated airway protection in patients with asthma is affected positively or negatively by propofol general anesthesia. The investigators hypothesized that the effects of propofol on asthmatic AMs and corresponding airway reactivity in vivo is different from the in vitro research. Through in vivo airway hyperresponsiveness (AHR) observation and clinical investigation of AM immune functions from asthma patients undergoing propofol general anesthesia to clarify the precise effects of propofol on AM immunity, and to provide theoretical basis for the clinical administration of propofol in asthmatic patients. This would optimize the practice of clinical anesthesia, especially for those with the tendency of AHR.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II;
* Aged from 18 years to 45 years;
* Patients with or without asthma or a history record of asthma;
* Undergoing elective lumpectomy under general anesthesia.

Exclusion Criteria:

* Allergy to propofol and opioids, a history of the use of centrally-acting drugs of any sort, chronic pain and psychiatric diseases records;
* Participants younger than 18yr，older than 45yr or pregnancy;
* Those who were not willing to or could not finish the whole study at any time;
* The PACU assessing score was under 6 on a scale of 10 (measuring somnolence, respiration, movement, color, and blood pressure on 0-2 scales), and arterial oxygen saturation measured by pulse oximetry (SaO2) was 92% or lower (supplemental oxygen was permitted).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with or without asthma undergoing general anesthesia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Alveolar macrophage viability assay | One day prior to the surgery, immediately after anaesthesia, at the beginning and the end of the operation and one day after surgeries.

SECONDARY OUTCOMES:
Alveolar macrophage phagocytosis Assay | One day prior to the surgery, immediately after anaesthesia, at the beginning and the end of the operation and one day after surgeries.
Alveolar macrophage cytokine Assay | One day before the surgery, immediately after anaesthesia, at the beginning and the end of the operation and one day after surgeries.
Mean airway pressure | Before operation to the end of the surgery.
Curve shape of CO2 | Before operation to the end of the surgery.
End-tidal CO2 | Before operation to the end of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China